CLINICAL TRIAL: NCT04843722
Title: Phase 1/2 Study of the Safety, Reactogenicity, and Immunogenicity of a Supplemental Spike & Nucleocapsid-targeted COVID-19 Vaccine to Enhance T Cell Based Immunogenicity in Participants Who Have Already Received Prime + Boost Vaccines Authorized For Emergency Use
Brief Title: COVID-19 Supplemental Vaccine Boost to Enhance T Cell Protection in Those Who Have Already Received EUA S-Based Vaccines
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The sponsor has changed the development plans which is not for safety reasons.
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: COVID-4.006
Record Dates: First submitted 2021-04-09; First posted 2021-04-13 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2021-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Open label 2 Cohort Phase 1 Study leading to Randomized Phase 2 Study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: hAd5-S-Fusion+N-ETSD at 5 × 10e10 IU/dose Subcutaneous (Experimental): Cohort 1 (n=20): hAd5-S-Fusion+N-ETSD at 5 × 10e10 IU/dose Subcutaneous on Day 1
  Interventions: Biological: hAd5-S-Fusion+N-ETSD vaccine
- Cohort 2: hAd5-S-Fusion+N-ETSD at 5 × 10e10 IU/dose Subcutaneous and 1 × 10e10 IU/dose Sublingual (Experimental): Cohort 2 (n=20): hAd5-S-Fusion+N-ETSD at 5 × 10e10 IU/dose Subcutaneous and 1 × 10e10 IU/dose Sublingual on Day 1
  Interventions: Biological: hAd5-S-Fusion+N-ETSD vaccine

INTERVENTIONS:
Biological: hAd5-S-Fusion+N-ETSD vaccine — Vaccine containing both full length wild type SARS-CoV-2 spike gene optimized for better spike protein expression, and full length wild type SARS-CoV-2 nucleocapsid gene modified to also contain an enhanced T cell stimulation domain (ETSD) to enhance cell-mediated immunity.

SUMMARY:
This is a phase 1/2 study in adult healthy subjects that have previously been vaccinated with an FDA-authorized vaccine against COVID-19. This clinical trial is designed to assess the safety, efficacy, reactogenicity, and immunogenicity of hAd5-S-Fusion+N-ETSD formulated for subcutaneous, sublingual, and oral (capsule) administration.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults, age ≥ 18 years, inclusive, at time of enrollment, that have previously received an FDA-authorized COVID-19 vaccine (both prime and boost) ≥14 days and

   ≤ 6 months before enrollment.
2. Able to understand and provide a signed informed consent that fulfills the relevant Institutional Review Board (IRB) or Independent Ethics Committee (IEC) guidelines.
3. Agrees to the collection of biospecimens (eg, NP swabs and/or saliva sample) and venous blood per protocol.
4. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
5. Ability to swallow a capsule.
6. Temperature < 38°C.
7. Agreement to practice effective contraception for female subjects of childbearing potential and non-sterile males. Female subjects of childbearing potential must agree to use effective contraception while on study until at least 1 month after the last dose of vaccine. Non-sterile male subjects must agree to use a condom while on study until at least 1 month after the last dose of vaccine. Effective contraception includes surgical sterilization (eg, vasectomy, tubal ligation), two forms of barrier methods (eg, condom, diaphragm) used with spermicide, IUDs, oral contraceptives, and abstinence.

Exclusion Criteria:

1. Persistent grade ≥ 2 AEs related to previous COVID-19 vaccination at the time of enrollment.
2. Allergy to any component of the investigational vaccine, or a more severe allergic reaction and history of allergies in the past.
3. Pregnant and nursing women. A negative serum or urine pregnancy test during screening and on the day of and prior to each dose must be documented before the vaccine is administered to a female subject of childbearing potential.
4. Chronic lung disease including chronic obstructive pulmonary disease (COPD) or moderate to severe asthma.
5. Pulmonary fibrosis.
6. Bone marrow or organ transplantation.
7. Extreme obesity (defined as BMI of 35 kg/m2 or higher).
8. Diabetes.
9. Chronic kidney disease.
10. Liver disease.
11. Sickle cell disease.
12. Thalassemia.
13. Any disease associated with acute fever, or any infection.
14. Self-reported history of SARS.
15. History of hepatitis B or hepatitis C.
16. HIV or other acquired or hereditary immunodeficiency.
17. Serious cardiovascular diseases, such as heart failure, coronary artery disease, cardiomyopathies, arrhythmia, conduction block, myocardial infarction, pulmonary hypertension, severe hypertension without controllable drugs, etc.
18. Cerebrovascular disease.
19. Cystic fibrosis.
20. Neurologic conditions, such as dementia.
21. Hereditary or acquired angioneurotic edema.
22. No spleen or functional asplenia.
23. Platelet disorder or other bleeding disorder that may cause injection contraindication.
24. Chronic use (more than 14 continuous days) of any medications that may be associated with impaired immune responsiveness within 3 months before administration of study vaccine. (Including, but not limited to, systemic corticosteroids exceeding 10 mg/day of prednisone equivalent, allergy injections, immunoglobulin, interferon, immunomodulators. The use of low dose topical, ophthalmic, inhaled and intranasal steroid preparations will be permitted.)
25. Prior administration of blood products in last 4 months.
26. Currently receiving treatment for cancer or history of cancer in the last five years (except basal cell carcinoma of the skin and cervical carcinoma in situ).
27. According to the judgement of investigator, various medical, psychological, social or other conditions that could affect the subjects ability to sign informed consent.
28. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Phase 1 Safety: Incidence of MAAEs and SAEs | through 1 week post final vaccine administration
  Incidence of MAAEs and SAEs through 1 week post final vaccine administration
Phase 1 Safety: Incidence and severity of solicited local reactogenicity AEs | through 1 week post final vaccine administration
  Incidence and severity of solicited local reactogenicity AEs through 1 week post final vaccine administration
Phase 1 Safety: Incidence and severity of solicited systemic reactogenicity AEs | through 1 week post final vaccine administration
  Incidence and severity of solicited systemic reactogenicity AEs through 1 week post final vaccine administration
Phase 1 Safety: Incidence and severity of unsolicited AEs | through 1 week post final vaccine administration
  Incidence and severity of unsolicited AEs through 1 week post final vaccine administration
Phase 1 Safety: Incidence of MAAEs and SAEs | through 30 days and 6 months post final vaccine administration
  Incidence of MAAEs and SAEs through 30 days and 6 months post final vaccine administration
Phase 1 Safety: Incidence and severity of unsolicited AEs | through 30 days post final vaccine administration
  Incidence and severity of unsolicited AEs through 30 days post final vaccine administration
Phase 1 Safety: Incidence of changes of laboratory safety examinations | Day 365
  Incidence of abnormal changes of laboratory safety examinations
Phase 1 Safety: Vital Sign - Temperature | Day 365
  Changes in vital signs from Grades 1-4:
  measured in (°C) or (°F)
Phase 1 Safety: Vital Sign - Heart Rate | Day 365
  Changes in vital signs from Grades 1-4:
  measured by how many heart beats per minute
Phase 1 Safety: Vital Sign - Blood Pressure | Day 365
  Changes in vital signs from Grades 1-4:
  systolic/diastolic - measured in mm Hg
Phase 1 Safety: Vital Sign - Respiratory Rate | Day 365
  Changes in vital signs from Grades 1-4:
  measured in how many breaths per minute
Phase 2 Efficacy: Percent of subjects that show an increase in N-reactive T cells | from baseline to Day 365
  Percent of subjects that show an increase in N-reactive T cells as assayed by N-Tiferon assay (≥ 25 pg/mL increase in cytokine concentration from baseline)

SECONDARY OUTCOMES:
Phase 1 Humoral Immunogenicity: GMT of S-specific and N-specific antibodies | Day 365
  GMT of S-specific and N-specific antibodies against 2019 novel coronavirus
Phase 1 Humoral Immunogenicity: GMT of neutralizing antibody | Day 365
  GMT of neutralizing antibody
Phase 1 Mucosal Immunogenicity: GMT of IgA antibody levels | Day 365
  GMT of IgA antibody levels
Phase 1 Cellular Immunogenicity: T cell activity | Day 365
  T cell activity against SARS-CoV-2 S protein and N protein. ImmunityBio has developed a rapid assay (N-Tiferon) to detect SARS-CoV-2-specific T cell responses directly in whole blood from participants in QUILT-4.001 vaccinated with hAd5 S-Fusion+N-ETSD targeting the S and N antigens of SARS-CoV-2. This assay detected interferon-γ (IFN-γ)-secreting S- and N-specific T cells directly in whole blood post-vaccination.
Phase 2 Efficacy: Incidence and severity of COVID-19 ≥14 days after vaccination | ≥14 days after vaccination
  Incidence and severity of COVID-19 ≥14 days after vaccination in subjects with no evidence of past SARS-CoV-2 infection. It applies to ≥3 for injection site reaction, fever, and other AEs. It also includes signs and symptoms of hypersensitivity which may include red rash (excluding site of injection), swollen throat or swollen areas of the body, wheezing, fainting, chest tightness, difficulty breathing, hoarse voice, difficulty swallowing, vomiting, diarrhea, and stomach cramping.
Phase 2 Efficacy: Mean SARS-CoV-2 viral load | Day 365
  Mean SARS-CoV-2 viral load for subjects with confirmed COVID-19 ≥14 days after vaccination
Phase 2 Efficacy: Humoral Immunogenicity - GMT of S-specific and N-specific antibodies | Day 365
  GMT of S-specific and N-specific antibodies against 2019 novel coronavirus
Phase 2 Efficacy: Humoral Immunogenicity - GMT of neutralizing antibody | Day 365
  GMT of neutralizing antibody
Phase 2 Efficacy: Mucosal Immunogenicity - GMT of IgA antibody levels | Day 365
  GMT of IgA antibody levels
Phase 2 Efficacy: Cellular Immunogenicity - T cell activity | Day 365
  T cell activity against SARS-CoV-2 S protein and N protein measured
Phase 2 Safety: Incidence of MAAEs and SAEs | through 1 week post final vaccine administration
  Incidence of MAAEs and SAEs through 1 week post final vaccine administration
Phase 2 Safety: Incidence and severity of solicited local reactogenicity AEs | through 1 week post final vaccine administration
  Incidence and severity of solicited local reactogenicity AEs through 1 week post final vaccine administration
Phase 2 Safety: Incidence and severity of solicited systemic reactogenicity AEs | through 1 week post final vaccine administration
  Incidence and severity of solicited systemic reactogenicity AEs through 1 week post final vaccine administration
Phase 2 Safety: Incidence and severity of unsolicited AEs | through 1 week post final vaccine administration
  Incidence and severity of unsolicited AEs through 1 week post final vaccine administration
Phase 2 Safety: Incidence of MAAEs and SAEs | through 30 days and 6 months post final vaccine administration
  Incidence of MAAEs and SAEs through 30 days and 6 months post final vaccine administration
Phase 2 Safety: Incidence and severity of unsolicited AEs | through 30 days post final vaccine administration
  Incidence and severity of unsolicited AEs through 30 days post final vaccine administration
Phase 2 Safety: Incidence of changes of laboratory safety examinations | Day 365
  Incidence of abnormal changes of laboratory safety examinations
Phase 2 Safety: Vital Sign - Temperature | Day 365
  Changes in vital signs from Grades 1-4:
  measured in (°C) or (°F)
Phase 2 Safety: Vital Sign - Heart rate | Day 365
  Changes in vital signs from Grades 1-4:
  measured by how many heart beats per minute
Phase 2 Safety: Vital Sign - Blood Pressure | Day 365
  Changes in vital signs from Grades 1-4:
  systolic/diastolic - measured in mm Hg
Phase 2 Safety: Vital Sign - Respiratory rate | Day 365
  Changes in vital signs from Grades 1-4:
  measured in how many breaths per minute

IPD SHARING:
Plan to Share IPD: No